CLINICAL TRIAL: NCT07081074
Title: ROS-scavenging Amino Acid-derived Lipids for the Prevention and Treatment of Radiation Dermatitis in Patients With Head and Neck Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024-134-3
Record Dates: First submitted 2025-07-15; First posted 2025-07-23 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-07

CONDITIONS: Radiation Dermatitis
MeSH Terms: conditions — Radiodermatitis | interventions — Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amino acid-derived lipids (Experimental)
  Interventions: Drug: Amino acid-derived lipids
- standard of care (Active Comparator)
  Interventions: Behavioral: standard of care

INTERVENTIONS:
Drug: Amino acid-derived lipids — Amino acid-derived lipids are applied to the treatment area, once daily during radiotherapy.
  Arms: Amino acid-derived lipids
Behavioral: standard of care — Standard of care
  Arms: standard of care

SUMMARY:
Radiation dermatitis is a common complication in head and neck squamous cell carcinoma patients receiving radiotherapy. This study proposes an ROS-scavenging amino acid-based nanolipid to prevent oxidative skin damage. A multicenter randomized trial will evaluate its safety and efficacy in reducing dermatitis severity and improving treatment continuity.

DETAILED DESCRIPTION:
Radiation dermatitis represents one of the most frequent complications in patients with head and neck squamous cell carcinoma (including nasopharyngeal carcinoma) undergoing radiotherapy, often leading to treatment interruption and compromised therapeutic outcomes. To address the limitations of current preventive strategies, this project proposes a novel amino acid-based lipid formulation designed to scavenge reactive oxygen species (ROS). Leveraging FDA-approved natural amino acids and engineered into a unique nanoliposomal structure, this formulation enables efficient delivery of antioxidative agents, effectively neutralizing excess ROS generated during radiotherapy while activating endogenous antioxidant signaling pathways, thereby mitigating oxidative damage to dermal cells. A multicenter randomized controlled clinical trial will be conducted to systematically evaluate the efficacy and safety of this intervention in reducing the incidence and severity of radiation dermatitis. This study will provide a clinically viable and safe prophylactic strategy, enhancing patients' quality of life and ensuring uninterrupted radiotherapy, with significant translational and societal implications.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a pathological diagnosis of non-metastatic head and neck malignant tumors;
2. Patients deemed suitable for high-dose radiotherapy, either as a primary treatment or as postoperative treatment following surgical resection.

Exclusion Criteria:

1. Eastern Cooperative Oncology Group performance status of >2;
2. Pre-existing skin rash, ulceration or open wound in the treatment area;
3. Known allergy to trolamine or amino acid;
4. Inflammatory or connective tissue disorder of the skin;
5. History of head and neck radiotherapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2025-09-23 (Estimated); Study Completion 2025-11-23 (Estimated)

PRIMARY OUTCOMES:
The incidence of radiation dermatitis | From the start of radiotherapy to 2 weeks after completion of radiotherapy.
  Patients are assessed weekly for radiation dermatitis by an experienced radiation oncology nurse according to the Radiation Therapy Oncology Group (RTOG) criteria.

SECONDARY OUTCOMES:
The maximum skin toxicity | From the start of radiotherapy to 2 weeks after completion of radiotherapy.
  The maximum grade of RTOG skin toxicity between 0 and 4.

CONTACTS AND LOCATIONS:
Overall Officials: Xingchen Peng, Principal Investigator — Sichuan University West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No